CLINICAL TRIAL: NCT05456412
Title: Influence of JAK Inhibitors on the Disease-associated Network of Intestinal Immune Cells in Ulcerative Colitis
Brief Title: JAK Inhibition in Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Galapagos NV (Industry)
Responsible Party: Principal Investigator, Andrea E. van der Meulen - de Jong, MD, PhD, Principal Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 81808
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Colitis, Ulcerative
Keywords: Janus Kinase Inhibitors
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Clinical practice protocol is followed. Additional biopsies and blood samples are taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment JAK inhibitor (Experimental): Clinical practice is followed for all patients treated with JAK inhibitor. Additional biopsies and blood is taken.
  Interventions: Other: JAK inhibitor treatment

INTERVENTIONS:
Other: JAK inhibitor treatment — Standard care

SUMMARY:
The treatment for Ulcerative Colitis (UC) aims to achieve and maintain remission and is usually lifelong and expensive. Current available medications are unable to break the cycle of chronic inflammation, and still a significant proportion of patients will fail to respond (primary non-response) or lose response over time (secondary non-response). There is now growing evidence that there is substantial interpatient variation in the composition of the inflammation associated network of immune cells. A deeper knowledge of the patient's alterations in the mucosal immune response would help identify key drivers of inflammation and select the appropriate therapy. By analyzing the changes in the composition of immune cells induced by Janus Kinase (JAK) inhibition, we aim to obtain a better insight into the mechanistic effects of JAK inhibition and the downstream effects. These mechanistic insights are needed to identifying potential responders and non-responders in the future.

ELIGIBILITY:
Age Ulcerative colitis active disease

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Multi-omics analyses of changes observed after JAK inhibition | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andrea van der Meulen, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided